CLINICAL TRIAL: NCT01361100
Title: Evaluation of the Oncoral® Test in Epidermoid Carcinomas of the Upper Aerodigestive Tract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Collaborators: Clinident Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ONCORAL; ET 2010-015 (Registry Identifier: Sponsor's number)
Record Dates: First submitted 2011-03-08; First posted 2011-05-26 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Carcinoma
Keywords: Otolaryngology
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oncoral test (Experimental)
  Interventions: Device: Oncoral® test

INTERVENTIONS:
Device: Oncoral® test — The patient rinses his oral cavity for 2 minutes. Then he screws lid back onto a beaker. The investigator holds the beaker straight so that the end of the aspiration mouth is dipped into the liquid. Then, the investigators takes 2 tubes and pushes them one after the other down on the opening of the beaker. The tubes should fill by themselves. The tubes can't be kept more than eleven days and are send to the Clinident Institute for the analysis.

SUMMARY:
This is a multicentric feasibility study aimed to evaluate the Oncoral® test. The study includes 2 steps. The first one aims to validate the algorithm defined at the time when the test was developed in patients with different tumour stages. Patients will be enrolled before any treatment. They will immediately undergo the test. No follow-up will be realized. In total, 100 patients will be included in this first step. The estimated period of inclusion is 6 months.

If the algorithm is validated, the second step of the study will start. The purpose is to determine the characteristics of the test. Enrollment will concern smokers and alcohol drinkers at high risk of developing an epidermoid carcinoma of the upper aerodigestive tract. Patient follow-up will vary with both the result of the test and the biopsy, up to a maximum of one year. In total, 385 patients will be enrolled in this step during an estimated period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

First step:

* Man or woman aged more than 40 years
* With frequent alcohol intoxication and/or smoking
* With histologically confirmed epidermoid carcinoma of the upper aerodigestive tract
* No treatment delivered for this disease
* Signed, written informed consent
* Mandatory affiliation with a health insurance system

Second step:

* Man or woman aged more than 40 years
* With frequent alcohol intoxication and/or smoking
* With no sign of an epidermoid carcinoma of the upper aerodigestive tract
* Signed, written informed consent
* Mandatory affiliation with a health insurance system

Exclusion Criteria:

First step:

* Previous history of cancer except carcinoma in situ of the uterine cervix or skin basal cell carcinoma treated with curative intent
* Gingivorrhagia when the test is realised
* Hypersensitivity to aspirin or to benzoate
* Asthmatic, diabetic patients or patents with chronic bronchitis requiring oxygen therapy
* Patients taking antibiotics at enrolment or during the previous week

Second step:

* Previous history of cancer except carcinoma in situ of the uterine cervix or skin basal cell carcinoma treated with curative intent
* Patient already treated for a cancer
* Gingivorrhagia when the test is realised
* Hypersensitivity to aspirin or to benzoate
* Asthmatic, diabetic patients or patients with chronic bronchitis requiring oxygen therapy
* Patients on antibiotics at enrolment or during the previous week

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Estimated)
Dates: Start 2010-12; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
First step: Confirm that the parameters used for the development of the test to qualify it as positive or negative lead to the same level of sensitivity (98%) | 1 year after the beginning of enrollment
  The algorithm was first defined when the test was developed in patients on different tumour stages .
Second step: Determine the characteristics of the Oncoral® test | 2 years after the beginning of the second step enrolment
  Sensitivity, specificity, positive predictive value, negative predictive value.

SECONDARY OUTCOMES:
First step: Estimation of test sensitivity | 1 year after the beginning of enrolment
  Sensitivity will be assessed by the calculation : true positives / (true positives + false negatives)
Second step : Estimation of test feasibility | 2 years after the beginning of the second step enrolment
  Feasibility will be assessed by :
  * the rate of patients who were not able to realise the test (difficulty to rinse the oral cavity)
  * the rate of tests that cannot be analysed (inadequate tests, problems of stability, difficulties with the extraction of volatile molecules, DNA or mRNA...) If the rate of unusable tests is greater than 10%, corrective actions will be necessary in order to use this test in the future. These actions will be considered according to the type of problems (adjustments of the test, transport...)
Second step: Estimation of the prevalence of epidermoid carcinoma of the upper aerodigestive tract in the target population | 3 years after the beginning of the second step enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ZROUNBA, MD, Principal Investigator — Centre Leon Berard
Locations (8):
- France (8):
  - CHU Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - CHU Caen Cote de Nacre, Caen
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Groupement Hospitalier Pitié Salpêtrière, Paris
  - Institut Curie, Paris
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Castellsague X, Quintana MJ, Martinez MC, Nieto A, Sanchez MJ, Juan A, Monner A, Carrera M, Agudo A, Quer M, Munoz N, Herrero R, Franceschi S, Bosch FX. The role of type of tobacco and type of alcoholic beverage in oral carcinogenesis. Int J Cancer. 2004 Feb 20;108(5):741-9. doi: 10.1002/ijc.11627. PMID 14696101
- [Background] Lingen MW, Kalmar JR, Karrison T, Speight PM. Critical evaluation of diagnostic aids for the detection of oral cancer. Oral Oncol. 2008 Jan;44(1):10-22. doi: 10.1016/j.oraloncology.2007.06.011. Epub 2007 Sep 6. PMID 17825602
- [Background] Nagler R, Bahar G, Shpitzer T, Feinmesser R. Concomitant analysis of salivary tumor markers--a new diagnostic tool for oral cancer. Clin Cancer Res. 2006 Jul 1;12(13):3979-84. doi: 10.1158/1078-0432.CCR-05-2412. PMID 16818695
- [Background] Tavassoli M, Brunel N, Maher R, Johnson NW, Soussi T. p53 antibodies in the saliva of patients with squamous cell carcinoma of the oral cavity. Int J Cancer. 1998 Oct 29;78(3):390-1. doi: 10.1002/(SICI)1097-0215(19981029)78:33.0.CO;2-9. No abstract available. PMID 9766578
- [Background] Peng G, Hakim M, Broza YY, Billan S, Abdah-Bortnyak R, Kuten A, Tisch U, Haick H. Detection of lung, breast, colorectal, and prostate cancers from exhaled breath using a single array of nanosensors. Br J Cancer. 2010 Aug 10;103(4):542-51. doi: 10.1038/sj.bjc.6605810. Epub 2010 Jul 20. PMID 20648015
- [Background] Mager DL, Haffajee AD, Devlin PM, Norris CM, Posner MR, Goodson JM. The salivary microbiota as a diagnostic indicator of oral cancer: a descriptive, non-randomized study of cancer-free and oral squamous cell carcinoma subjects. J Transl Med. 2005 Jul 7;3:27. doi: 10.1186/1479-5876-3-27. PMID 15987522
- [Background] Li Y, St John MA, Zhou X, Kim Y, Sinha U, Jordan RC, Eisele D, Abemayor E, Elashoff D, Park NH, Wong DT. Salivary transcriptome diagnostics for oral cancer detection. Clin Cancer Res. 2004 Dec 15;10(24):8442-50. doi: 10.1158/1078-0432.CCR-04-1167. PMID 15623624
- [Background] El-Naggar AK, Mao L, Staerkel G, Coombes MM, Tucker SL, Luna MA, Clayman GL, Lippman S, Goepfert H. Genetic heterogeneity in saliva from patients with oral squamous carcinomas: implications in molecular diagnosis and screening. J Mol Diagn. 2001 Nov;3(4):164-70. doi: 10.1016/S1525-1578(10)60668-X. PMID 11687600
- [Background] Liao PH, Chang YC, Huang MF, Tai KW, Chou MY. Mutation of p53 gene codon 63 in saliva as a molecular marker for oral squamous cell carcinomas. Oral Oncol. 2000 May;36(3):272-6. doi: 10.1016/s1368-8375(00)00005-1. PMID 10793330
- [Background] Anker P, Lyautey J, Lederrey C, Stroun M. Circulating nucleic acids in plasma or serum. Clin Chim Acta. 2001 Nov;313(1-2):143-6. doi: 10.1016/s0009-8981(01)00666-0. PMID 11694252
- [Background] Li Y, Zhou X, St John MA, Wong DT. RNA profiling of cell-free saliva using microarray technology. J Dent Res. 2004 Mar;83(3):199-203. doi: 10.1177/154405910408300303. PMID 14981119
- [Background] Rieger-Christ KM, Mourtzinos A, Lee PJ, Zagha RM, Cain J, Silverman M, Libertino JA, Summerhayes IC. Identification of fibroblast growth factor receptor 3 mutations in urine sediment DNA samples complements cytology in bladder tumor detection. Cancer. 2003 Aug 15;98(4):737-44. doi: 10.1002/cncr.11536. PMID 12910517
- [Background] Phillips M, Gleeson K, Hughes JM, Greenberg J, Cataneo RN, Baker L, McVay WP. Volatile organic compounds in breath as markers of lung cancer: a cross-sectional study. Lancet. 1999 Jun 5;353(9168):1930-3. doi: 10.1016/S0140-6736(98)07552-7. PMID 10371572
- [Background] Miekisch W, Schubert JK, Noeldge-Schomburg GF. Diagnostic potential of breath analysis--focus on volatile organic compounds. Clin Chim Acta. 2004 Sep;347(1-2):25-39. doi: 10.1016/j.cccn.2004.04.023. PMID 15313139